CLINICAL TRIAL: NCT03994861
Title: Validation and Reliability of the Dutch Version of the Fear-Avoidance Component Scale (FACS)
Brief Title: Dutch Version Fear-Avoidance Component Scale (FACS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Lotte Janssens, Prof. dr., Hasselt University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 18.61/REVA18.02
Record Dates: First submitted 2019-06-04; First posted 2019-06-21 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Musculoskeletal Pain; Musculoskeletal Pain Disorder; Fear of Pain; Fear of Injury; Low Back Pain, Recurrent; Neck Pain; Shoulder Pain; Knee Pain Chronic; Hip Pain Chronic; PROMs
MeSH Terms: conditions — Musculoskeletal Pain; Collagen Diseases; Low Back Pain; Neck Pain; Shoulder Pain

STUDY DESIGN:
Intervention Model Description: Patients with musculoskeletal disorders are compared to matched healthy controls.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with musculoskeletal disorders (Active Comparator): Patients with either shoulder pain, knee pain, hip pain, low back pain, pelvic pain or neck pain as their primary pain complaint, lasting for 6 weeks or longer
  Interventions: Diagnostic Test: Assessment of disability and behavior (by questionnaires)
- Healthy controls (Sham Comparator): Age- and gender-matched healthy controls (without musculoskeletal pain)
  Interventions: Diagnostic Test: Assessment of disability and behavior (by questionnaires)

INTERVENTIONS:
Diagnostic Test: Assessment of disability and behavior (by questionnaires) — Assessment of disability and behavior (by questionnaires)

SUMMARY:
Chronic musculoskeletal disorders such as low back and neck pain are responsible for an enormous global burden. Fear-avoidance (FA) can be a predictor for the transition from subacute to chronic low back pain. In patients with neck pain, those who were less fearful about harming their neck, had higher pain tolerance, which might have a positive impact on their level of disability. A new scale, the Fear-Avoidance Component Scale (FACS) was developed by Neblett, Mayer, Hartzell, Williams and Gatchel (2015) to assess FA. It consists of an all-encompassing set of constructs that more effectively deals with all critical issues of the FA concept than current scales do. Current scales have been criticized because of following findings: limited construct validity, little evidence on treatment responsiveness, a lack of evidence-based cut-off scores and items being too narrow or too general. The new scale comprehensively assesses all cognitive, emotional and behavioral components related to the updated version of the FA model by combining items of well-known scales in context of the FA model with items on one's perception of victimization and blame related to an injury. A Dutch version of the FACS is currently lacking. Subsequently, the aim of this study is to investigate different psychometric properties of the generated Dutch version in patients with musculoskeletal disorders.

ELIGIBILITY:
Inclusion criteria for all patients

* between 18-80 years old
* current pain complaint is not surgically treated
* not being currently treated by a physiotherapist for pain complaint
* Dutch language is mother tongue
* At least 6 weeks of pain Exclusion criteria for all patients
* Pain from a non-musculoskeletal origin (e.g., tumour)
* neurological disease
* impaired cognition Inclusion criteria for healthy controls
* Not being disabled due to MSK pain based on cut-off per disability questionnaire
* Between 18-80 years old
* Dutch language is mother tongue

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
The fear-avoidance component scale (FACS) | day 0
  Questionnaire evaluating fear-avoidance related to pain (for all participants) 20 items range from 0-100
The fear-avoidance component scale (FACS) | day 7
  Questionnaire evaluating fear-avoidance related to pain (for all participants) 20 items range from 0-100
Disabilities of the arm, shoulder and hand questionnaire (DASH) for shoulder pain patients | day 0
  Questionnaire evaluating disability (only used in patients with shoulder pain) 30 items Range total score 0-100 5 point-scale
Disabilities of the arm, shoulder and hand questionnaire (DASH) for shoulder pain patients | day 7
  Questionnaire evaluating disability (only used in patients with shoulder pain) 30 items Range total score 0-100 5 point-scale
Hip disability and Osteoarthritis Outcome Score (HOOS) for hip pain patients | day 0
  Questionnaire evaluating disability (only used in patients with hip pain) Subscores per domain 40 items 5 point scale 5 domains: symptoms (5 items), pain (10 items), activities of daily living (17 items), sport and leisure time (4 items), quality of life (4 items)
Hip disability and Osteoarthritis Outcome Score (HOOS) for hip pain patients | day 7
  Questionnaire evaluating disability (only used in patients with hip pain) Subscores per domain 40 items 5 point scale 5 domains: symptoms (5 items), pain (10 items), activities of daily living (17 items), sport and leisure time (4 items), quality of life (4 items)
Knee injury and Osteoarthritis Outcome Score (KOOS) for knee pain patients | day 0
  Questionnaire evaluating disability (only used in patients with knee pain) Subscores per domain 42 items 5 domains: pain (9 items), symptoms (7 items), activities of daily life (17 items), sports and leisure (5 items), quality of life (4 items) 5 point Likert scale
Knee injury and Osteoarthritis Outcome Score (KOOS) for knee pain patients | day 7
  Questionnaire evaluating disability (only used in patients with knee pain) Subscores per domain 42 items 5 domains: pain (9 items), symptoms (7 items), activities of daily life (17 items), sports and leisure (5 items), quality of life (4 items) 5 point Likert scale
Oswestry Disability Index for patients with low back pain | day 0
  Questionnaire evaluating disability (only used in patients with low back pain) 10 items Total score range from 0-100
Oswestry Disability Index for patients with low back pain | day 7
  Questionnaire evaluating disability (only used in patients with low back pain) 10 items Total score range from 0-100
Neck Disability Index for neck pain patients | day 0
  Questionnaire evaluating disability (only used in patients with neck pain) 10 items Total score range from 0-100
Neck Disability Index for neck pain patients | day 7
  Questionnaire evaluating disability (only used in patients with neck pain) 10 items Total score range from 0-100
Fear-avoidance beliefs questionnaire | day 0
  3 subscales: physical activity (4 items; 0-30), work (7 items; 0-66) and rest (5 items)
Fear-avoidance beliefs questionnaire | day 7
  3 subscales: physical activity (4 items; 0-30), work (7 items; 0-66) and rest (5 items)
Tampa scale for kinesiophobia | day 0
  Questionnaire evaluating kinesiophobia related to pain (for all participants) 17 items total score from 17-68
Tampa scale for kinesiophobia | day 7
  Questionnaire evaluating kinesiophobia related to pain (for all participants) 17 items total score from 17-68
Pain catastrophizing scale | day 0
  Questionnaire evaluating catastrophizing (for all participants) 13 items 5 point Likert Scale Total score 0-52
Pain catastrophizing scale | day 7
  Questionnaire evaluating catastrophizing (for all participants) 13 items 5 point Likert Scale Total score 0-52
IEQ-Dutch scale for perceived injustice | day 0
  Questionnaire evaluating perceived injustice (for all participants) 12 items 5 point Likert-scale Total score range 0-48
IEQ-Dutch scale for perceived injustice | day 7
  Questionnaire evaluating perceived injustice (for all participants) 12 items 5 point Likert-scale Total score range 0-48
Hospital anxiety and depression scale | day 0
  Questionnaire evaluating anxiety and depression (for all participants) 2 subscales: anxiety (7 items) and depression (7 items) Total score 0-21 per subscale
Hospital anxiety and depression scale | day 7
  Questionnaire evaluating anxiety and depression (for all participants) 2 subscales: anxiety (7 items) and depression (7 items) Total score 0-21 per subscale

CONTACTS AND LOCATIONS:
Overall Officials: Annick Timmermans, PhD, PT, Principal Investigator — Hasselt University
Locations (1):
- Lotte Janssens, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: No